CLINICAL TRIAL: NCT01751932
Title: Standardized Procedure for the Assessment of New-to-market Continuous Glucose Monitoring Systems
Acronym: SPACE2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.H. DeVries, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPACE2
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Last update posted 2013-12-16 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CGM Monitoring (Experimental): Fitting of Dexcom G4 Platinum CGM monitor and Medtronic Enlite CGM monitor
  Interventions: Device: CGM Monitoring

INTERVENTIONS:
Device: CGM Monitoring — All patients will be fitted with the two study CGM systems. Paradigm Veo will be configured to use the CGM part only if another pump is used.
  Other Names: Dexcom G4 Platinum and Medtronic Enlite CGM

SUMMARY:
The purpose of this study is to assess the accuracy of two continuous glucose monitoring devices (the Dexcom G4 Platinum and Medtronic Enlite systems) in patients with type 1 diabetes mellitus.

DETAILED DESCRIPTION:
The study will use two CE marked Continuous Glucose Monitoring (CGM) systems; Dexcom G4 Platinum CGM CE-marked 2012 (Dexcom, USA) and the Medtronic Paradigm Veo system with Enlite Sensor CE-marked 2011 (Medtronic, USA). Both the Dexcom G4 Platinum and the Medtronic Enlite sensors will be obtained through normal commercial channels rather than directly from the manufacturer. The two CGM sensors will be worn concomitantly by the participant during the visit to the Clinical Research Center (CRC). This visit will have a duration of 6 hours. Blood will be drawn for the determination of glucose levels. The patient will receive his usual breakfast and an increased insulin bolus (180% of the patient's calculated mealtime dose) will be administered to correct the breakfast glucose excursion with the aim of inducing a period of minor hypoglycaemia. Blood sampling will continue until the end of the admission. At the end of this CRC part, the patient will continue to wear the two sensors at home. In the case of sensor failure before the CRC session on the third day into the study, patients will be instructed to insert a new sensor per the manufacturer's instruction for use and to notify study coordinators of the event. Sensors will be worn until the end of the six day study duration. Patients will be asked to perform at least 6 fingersticks per day for blood glucose measurements with the study glucometer. The study will end on the 6th day after initial sensor insertion. Patients will return to the CRC to have the sensor removed and their CGM sensor and blood glucometer data downloaded from the devices. In case of failure of both sensors after the CRC session but before the scheduled six day study duration, patients will return to the CRC for sensor removal and for data download.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* diagnosed with Type 1 diabetes mellitus at least 6 months according to the WHO definition
* Body Mass Index (BMI) <35 kg/m²
* willing and able to wear a CGM device for the duration of the study and undergo all study procedures
* HbA1c <10%
* signed informed consent form prior to study entry

Exclusion Criteria:

* Patient is pregnant, or breast feeding during the period of the study.
* Patient is using a medication that significantly impacts glucose metabolism (oral steroids) except if stable for at least the last three months and expected to remain stable for the study duration
* Patient may not use acetaminophen (paracetamol) while participating in the study
* Has severe medical or psychological condition(s) or chronic conditions/infections that in the opinion of the Investigator would compromise the patient's safety or successful participation in the study.
* Patient is actively enrolled in another clinical trial or took part in a study within 30 days
* Known adrenal gland problem, pancreatic tumour, or insulinoma
* Inability of the patient to comply with all study procedures
* Inability of the patient to understand the patient information.
* Patient donated blood in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-01; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Mean Absolute Relative Difference (MARD) | up to day 6 of use
  MARD will be assessed as an average of the first 6 days of wear

SECONDARY OUTCOMES:
Accuracy of sensors per glycemic range and trial phase | up to day 6 of use
  Accuracy of the sensor in the hypoglycaemic (defined as a blood glucose value ≤3.9 mmol/L) and hyperglycaemic area (defined as a blood glucose value ≥10.0 mmol/L) as an average of the first six days of use. Additionally, a separate analysis will be performed to assess sensor performance and accuracy per day of sensor life.

CONTACTS AND LOCATIONS:
Overall Officials: J. Hans DeVries, MD, PhD, Principal Investigator — Academic Medical Center - Department of Internal Medicine, Amsterdam, The Netherlands; Eric Renard, PhD, Principal Investigator — Medical University Montpellier, France; Angelo Avogaro, PhD, Principal Investigator — Medical University Padova, Italy; Julia Mader, MD, Study Director — Medical University Graz, Austria; Thomas Pieber, MD, Principal Investigator — Medical University Graz, Austria
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Derived] Kropff J, Bruttomesso D, Doll W, Farret A, Galasso S, Luijf YM, Mader JK, Place J, Boscari F, Pieber TR, Renard E, DeVries JH. Accuracy of two continuous glucose monitoring systems: a head-to-head comparison under clinical research centre and daily life conditions. Diabetes Obes Metab. 2015 Apr;17(4):343-9. doi: 10.1111/dom.12378. Epub 2014 Sep 10. PMID 25132320